CLINICAL TRIAL: NCT00656890
Title: A Phase 2, Multi-dose, Double-blind, Placebo-controlled, Randomized, Multicenter Study of MDX-1100 (Anti-CXCL10 Human Monoclonal Antibody) in Subjects With Active Ulcerative Colitis
Brief Title: A Study of MDX-1100 in Subjects With Active Ulcerative Colitis
Acronym: MDX1100-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDX1100-06; IM129-004 (Other: BMS)
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis, rectal bleeding
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Hemorrhage | interventions — Injections; MDX-1100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): sterile saline for injection
  Interventions: Biological: sterile saline for injection
- 1 (Experimental): MDX-1100 for injection
  Interventions: Biological: MDX-1100

INTERVENTIONS:
Biological: sterile saline for injection — 10mg/kg/dose sterile saline injected every other week for a total of 4 doses
  Arms: 2
Biological: MDX-1100 — 10mg/kg/dose MDX-1100 injected every other week for a total of 4 doses
  Arms: 1

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the MDX-1100 regimen in subjects with active Ulcerative colitis(UC) and determine the response rate at day 57 in patients administered MDX-1100.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active UC on either 5-ASA,corticosteroids,azathioprine(AZA) and or/6-mercaptopurine(6-MP);
* Mayo score of 6 to 10 points with moderate to severe disease on endoscopy
* Subjects on the following medications;

  1. prednisolone ≤ 20 mg daily (or equivalent) (dose must be stable for at least 2 weeks prior to study drug administration)
  2. 5-ASA (dose must be stable for at least 4 weeks prior to study drug administration)
  3. AZA or 6-MP (dose must be stable for at least 3 months prior to study drug administration)
  4. Rectal steroids or 5-ASA (must have been stable for at least 4 weeks prior to study drug)

Exclusion Criteria:

* Anti-TNF therapy within 8 weeks before study drug administration
* Contraindication to colonoscopy or sigmoidoscopy
* Primary or secondary immunodeficiency
* Autoimmune disease besides UC, with the exceptions of Sjogren's syndrome or hypothyroidism
* History of malignancy, excluding adequately treated and cured basal or squamous cell of the skin, or cervical carcinoma in situ
* Evidence of acute or chronic infection
* Clinically significant disease requiring medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in Mayo score at Day 57 compared with Screening | Day 57

SECONDARY OUTCOMES:
the remission rate | Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (7):
  - Advanced Medical Research Center, Port Orange, Florida
  - Florida Medical Clinic-Tampa Clinic, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Dayton Science Institute, Dayton, Ohio
- Canada (3):
  - Abbotsford, British Columbia
  - Vancouver, British Columbia
  - Toronto, Ontario
- Czechia (6):
  - Olomouc
  - Prague
  - Strakonice
  - Tábor
  - Ústí nad Labem
  - Valasske Mezifici
- Hungary (9):
  - Budapest
  - Debrecen
  - Gyula
  - Kaposvár
  - Kecskemét
  - Nagykanizsa
  - Siófok
  - Vác
  - Zalaegerszeg
- Latvia (3):
  - Daugavpils
  - Riga
  - Valmiera
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Tg. Mures
  - Timișoara
- Russia (3):
  - Moscow
  - Saratov
  - Yaroslavl
- Ukraine (8):
  - Chernivtsy
  - Dniepropetrovsk
  - Donetsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Simferopol

REFERENCES:
- [Derived] Mayer L, Sandborn WJ, Stepanov Y, Geboes K, Hardi R, Yellin M, Tao X, Xu LA, Salter-Cid L, Gujrathi S, Aranda R, Luo AY. Anti-IP-10 antibody (BMS-936557) for ulcerative colitis: a phase II randomised study. Gut. 2014 Mar;63(3):442-50. doi: 10.1136/gutjnl-2012-303424. Epub 2013 Mar 5. PMID 23461895